CLINICAL TRIAL: NCT03671824
Title: The Difficult Airway: Incidence and Predictors in Lean vs. Obese Patients in a Large Public Teaching Hospital
Brief Title: The Difficult Airway
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Tiffany B Moon, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 022016-055
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Intubation;Difficult
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lean: BMI ≤ 30 kg/m2
  Interventions: Other: Measurements
- Obese: BMI ≥30 kg/m2
  Interventions: Other: Measurements

INTERVENTIONS:
Other: Measurements — Physiologic measurements including but not limited to thyromental distance, sternomental distance, Mallampati score, mouth opening, interincisor distance, and mandibular protrusion will be measured and recorded. All measurements are non invasive.

SUMMARY:
Patients who are obese, as defined by a BMI ≥ 30 kg/m2 may be more difficult to intubate than non-obese patients. Traditional methods of airway assessment such as Mallampati score, mouth opening, and thyromental distance may not be the best predictors of difficult intubation. Patients who are scheduled to have non-stat surgery at Parkland Memorial Hospital will be asked to participate in this study and sign a written consent form. Physiologic measurements including but not limited to thyromental distance, sternomental distance, Mallampati score, mouth opening, interincisor distance, and mandibular protrusion will be measured and recorded. All measurements are non invasive. The remaining aspects of perioperative care, including the general anesthetic technique, will be standardized for all patients and will not differ from the standard of care. There will be no incentive or payment to the patients. This prospective study is intended to enroll 4500 consecutive surgical patients. Lean patients (BMI < 30 kg/m2) who are intubated by the same anesthesia providers during the same time period will be included as the control group and to report the incidence of difficult mask ventilation and difficult intubation in our general surgical population, which has not previously been defined.

DETAILED DESCRIPTION:
The study will enroll 4500 ASA physical status 1-4 patients who are scheduled to undergo surgery under general endotracheal anesthesia (GETA) at Parkland Hospital. A research assistant will identify eligible patients using the electronic medical record. After it is deemed that the patient satisfies all inclusion and exclusion criteria, the anesthesia provider or research assistant will approach the patient in the preoperative surgery holding area to ask for their permission to enroll in the study. Only study team personnel will ask potential patients for participation in the study; anesthesia providers who are not study team personnel will not be allowed to consent patients for the study. All relevant information to the study will be provided and the patient will be asked to sign an informed consent. After consent is obtained, measurements of the patient's anatomical features including thyromental distance, sternomental distance, neck circumference, interincisor distance, mandibular protrusion, and Mallampati score will be taken and recorded by the research assistant or anesthesia provider.

In the operating room, patients will have standard ASA monitors (NIBP, SpO2, EKG, ETCO2, temperature) placed. Lean patients will be placed in the standard "sniffing" position while obese patients will be placed in the "ramped" position as previously described. All patients will undergo pre-oxygenation for at least 3 minutes prior to induction of anesthesia. Patients will undergo induction of general anesthesia according to a standardized protocol that does not differ from the usual standard of care. The initial blade used for laryngoscopy will be selected by the anesthesia provider according to the characteristics of the patient as has been recommended by previous authors. After induction of general anesthesia, a research assistant will ask the anesthesia provider the degree of difficulty of mask ventilation and laryngoscopy using a standardized questionnaire modified from the intubation difficulty score. For mask ventilation, any adjunct use of equipment such as an oral airway or nasopharyngeal airway will be recorded. If two-handed ventilation is used, it will be recorded as well. The type of laryngoscope blade and Cormack-Lehane grade during laryngoscopy will be recorded. The level of training of the laryngoscopist (resident vs CRNAs vs faculty) and how many years they have been in that role will be recorded. The time from induction to intubation will also be recorded, based on the time those events are marked in the electronic medical record, as well as the lowest SpO2 that occurred between induction to intubation.

The intubation difficulty scale (IDS), which has previously been validated, will be used to score the intubation. This scale has been used in comparing difficult tracheal intubation in lean vs. obese patients.

The IDS will be comprised of 7 questions with numerical values for each question, resulting in a cumulative score. Those with an IDS score <5 will be considered "not difficult" and those with an IDS score ≥5 will be considered "difficult." A "failed intubation" will be defined as that in which the airway cannot be secured in a non-invasive fashion (e.g., cricothyrotomy) or the patient has to be awakened. The 7 questioned used to determine the IDS score will be the same as those used by Adnet et al:

1. Number of additional intubation attempts
2. Number of additional operators
3. Number of alternative intubation techniques used
4. Laryngoscopic view (Grade 1 = 0, Grade 2 = 1, Grade 3 = 2, Grade 4 = 3)

   Cormack Lehane grades [13]:
   * Grade 1- vocal cords completely visible
   * Grade 2- arytenoids visible but cords not completely visible
   * Grade 3- only epiglottis visible
   * Grade 4- epiglottis not visible
5. Lifting force applied during laryngoscopy (0 if inconsiderable and 1 if considerable force used)
6. External laryngeal pressure applied for optimized glottic exposure (0 if no, 1 if yes)
7. Position of vocal cords at intubation (0 if abducted or not visible, 1 if adducted)

Protected patient information including name, medical record number, and date of birth will be recorded. Demographic data such as height, weight, BMI, race, and gender will also be recorded. All patients will receive a standardized general anesthetic that is usual and customary for patients undergoing their scheduled operation.

Additional information gathered will include ASA status, presence of comorbidities (e.g, OSA, HTN, DM), thyromental distance, sternomental distance, ability to protrude mandibular teeth over maxillary teeth, interincisor distance, ability to have full range of motion of the neck, Mallampati score, and neck circumference.

* Neck circumference will be measured at the level of the cricoid cartilage with the patient's neck in neutral position.
* Thyromental distance is thought to be an indicator of mandibular space. It will be measured as the distance from the prominentia laryngea of the thyroid cartilage to the symphysis of the mandible with the patient in maximum neck extension with the mouth closed.
* Sternomental distance will be measured as the distance from the sternal notch to the symphysis of the mandible with the patient in maximum neck extension with the mouth closed.
* Mallampati status will be obtained with the patient in an upright sitting position with the head in neutral position. Patients will be asked to open their mouth as wide as possible with tongue protrusion without phonation. Pharyngeal structures will be assess and classification will be performed according to the structures seen (Class 1 = soft palate, fauces, uvula, tonsillar pillars; Class 2 = soft palate, fauces, uvula; Class 3 = soft palate, base of uvula only; Class 4 = soft palate not visible).
* The ability of the patient to protrude their lower teeth over their upper lip (upper lip bite test) will be assessed. Class 1 = lower incisors can bite the upper lip above the vermilion line; Class 2 = lower incisors can bite the upper lip below the vermilion line; Class 3 = lower incisors cannot bite the upper lip [9].
* Neck range of motion will be graded on a binary scale. Those will full range of motion in flexion and extension will be graded as full and those without full range of motion will be graded as limited.
* Interincisor distance will be measured as the maximum distance between the central incisors (teeth 9 and 24 or teeth 8 and 25). Patients who are edentulous will have their gum-to-gum distance recorded as the interincisor distance.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* ASA physical status classification 1 to 4
* Scheduled for an operation that requires general endotracheal anesthesia
* Willing and able to consent in English or with use of appropriate language translator
* Anesthesia providers who are caring for patients who have enrolled in the study will also be potential subjects who will be verbally consented and asked to fill out a questionnaire.

Exclusion Criteria:

* Age less than 18 or older than 80
* Unable to give informed consent for participation in the study
* Stat cases
* Patients who will not be expected to have general anesthesia (e.g., monitored anesthesia care or regional anesthesia)
* Patient refusal
* History of difficult intubation
* Planned awake fiberoptic intubation
* Previous neck surgery (on bone, joint, or soft tissues in neck) or radiation
* Obvious neck pathology/abnormality

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to have non-stat surgery at Parkland Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 4022 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study will be the incidence of difficult mask ventilation and intubation in lean vs. obese patients. | Intraoperative
  Incidence of DI and DMV

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Moon, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Background] Braz LG, Braz DG, Cruz DS, Fernandes LA, Modolo NS, Braz JR. Mortality in anesthesia: a systematic review. Clinics (Sao Paulo). 2009;64(10):999-1006. doi: 10.1590/S1807-59322009001000011. PMID 19841708
- [Background] Brodsky JB, Lemmens HJ, Brock-Utne JG, Vierra M, Saidman LJ. Morbid obesity and tracheal intubation. Anesth Analg. 2002 Mar;94(3):732-6; table of contents. doi: 10.1097/00000539-200203000-00047. PMID 11867407
- [Background] Shiga T, Wajima Z, Inoue T, Sakamoto A. Predicting difficult intubation in apparently normal patients: a meta-analysis of bedside screening test performance. Anesthesiology. 2005 Aug;103(2):429-37. doi: 10.1097/00000542-200508000-00027. PMID 16052126
- [Background] Sturm R, Hattori A. Morbid obesity rates continue to rise rapidly in the United States. Int J Obes (Lond). 2013 Jun;37(6):889-91. doi: 10.1038/ijo.2012.159. PMID 22986681
- [Background] Benumof JL. Obstructive sleep apnea in the adult obese patient: implications for airway management. J Clin Anesth. 2001 Mar;13(2):144-56. doi: 10.1016/s0952-8180(01)00232-x. PMID 11331179
- [Background] Juvin P, Lavaut E, Dupont H, Lefevre P, Demetriou M, Dumoulin JL, Desmonts JM. Difficult tracheal intubation is more common in obese than in lean patients. Anesth Analg. 2003 Aug;97(2):595-600. doi: 10.1213/01.ANE.0000072547.75928.B0. PMID 12873960
- [Background] Neligan PJ, Porter S, Max B, Malhotra G, Greenblatt EP, Ochroch EA. Obstructive sleep apnea is not a risk factor for difficult intubation in morbidly obese patients. Anesth Analg. 2009 Oct;109(4):1182-6. doi: 10.1213/ane.0b013e3181b12a0c. PMID 19762747
- [Background] Khan ZH, Mohammadi M, Rasouli MR, Farrokhnia F, Khan RH. The diagnostic value of the upper lip bite test combined with sternomental distance, thyromental distance, and interincisor distance for prediction of easy laryngoscopy and intubation: a prospective study. Anesth Analg. 2009 Sep;109(3):822-4. doi: 10.1213/ane.0b013e3181af7f0d. PMID 19690252
- [Background] Turkan S, Ates Y, Cuhruk H, Tekdemir I. Should we reevaluate the variables for predicting the difficult airway in anesthesiology? Anesth Analg. 2002 May;94(5):1340-4, table of contents. doi: 10.1097/00000539-200205000-00055. PMID 11973217
- [Background] Collins JS, Lemmens HJ, Brodsky JB, Brock-Utne JG, Levitan RM. Laryngoscopy and morbid obesity: a comparison of the "sniff" and "ramped" positions. Obes Surg. 2004 Oct;14(9):1171-5. doi: 10.1381/0960892042386869. PMID 15527629
- [Background] Kim WH, Ahn HJ, Lee CJ, Shin BS, Ko JS, Choi SJ, Ryu SA. Neck circumference to thyromental distance ratio: a new predictor of difficult intubation in obese patients. Br J Anaesth. 2011 May;106(5):743-8. doi: 10.1093/bja/aer024. Epub 2011 Feb 24. PMID 21354999
- [Background] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827
- [Background] Al Ramadhani S, Mohamed LA, Rocke DA, Gouws E. Sternomental distance as the sole predictor of difficult laryngoscopy in obstetric anaesthesia. Br J Anaesth. 1996 Sep;77(3):312-6. doi: 10.1093/bja/77.3.312. PMID 8949801
- [Background] Mallampati SR, Gatt SP, Gugino LD, Desai SP, Waraksa B, Freiberger D, Liu PL. A clinical sign to predict difficult tracheal intubation: a prospective study. Can Anaesth Soc J. 1985 Jul;32(4):429-34. doi: 10.1007/BF03011357. PMID 4027773
- [Background] Sheff SR, May MC, Carlisle SE, Kallies KJ, Mathiason MA, Kothari SN. Predictors of a difficult intubation in the bariatric patient: does preoperative body mass index matter? Surg Obes Relat Dis. 2013 May-Jun;9(3):344-9. doi: 10.1016/j.soard.2012.02.004. Epub 2012 Mar 3. PMID 22475762
- [Background] Vittinghoff E, McCulloch CE. Relaxing the rule of ten events per variable in logistic and Cox regression. Am J Epidemiol. 2007 Mar 15;165(6):710-8. doi: 10.1093/aje/kwk052. Epub 2006 Dec 20. PMID 17182981